CLINICAL TRIAL: NCT02029508
Title: The Effectiveness Comparison of Three Different Methods for the Treatment of Posterior Semicircular Canal Benign Paroxysmal Positional Vertigo: Prospective, Double Blinded, Randomized, Multicenter Clinical Trial
Brief Title: The Treatment of Posterior Semicircular Canal Benign Paroxysmal Positional Vertigo
Acronym: BPPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hong Ju Park, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSCC_BPPV_Kr
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: PSCC(Posterior semicircular canal); BPPV(Bening paroxysmal positional vertigo); Vertigo; Otorhinolaryngologic Diseases
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Otorhinolaryngologic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Epley maneuver (Active Comparator): The group using modified Epley maneuver for PSCC BPPV
  Interventions: Procedure: Modified Epley maneuver
- Semont maneuver (Active Comparator): The group using Semont maneuver for PSCC BPPV
  Interventions: Procedure: Semont maneuver
- Sham (Sham Comparator): The group using Reverse Epley maneuver for PSCC BPPV
  Interventions: Procedure: Reverse Epley maneuver

INTERVENTIONS:
Procedure: Modified Epley maneuver — For Modified Epley maneuver, the patient was placed in the upright position with the head turned 45 degrees toward the affected ear. And then the patient was rapidly laid back to the supine head-hanging position for 1 minute. Next, the head was turned 90 degrees toward the other (unaffected) side for 1 minute. Next, the head is turned a further 90 degrees (usually necessitating the patient's body to also move from the supine position to the lateral decubitus position) such that the patient' head is nearly in the facedown position for 1 minute. The patient is then brought into the upright sitting position for 1 minute, completing the maneuver.
  Arms: Epley maneuver
Procedure: Semont maneuver — Patient's head was turned 45 degrees toward the healthy side. And then patient was rapidly moved to affected side-lying position and sustained for 2 minutes. Next, Patient is rapidly taken to the opposite side-lying position without pausing in the sitting position or changing the head position relative to the shoulder for 2 minutes. Next, Patient returns slowly with the head still tilted and fixed until the seated position for 1 minute.
  Arms: Semont maneuver
Procedure: Reverse Epley maneuver — Like the modified Epley maneuver, but the direction was reverse.
  Arms: Sham

SUMMARY:
The purpose of this study was to compare the treatment effectiveness of three different methods for posterior semicircular canal benign paroxysmal positional vertigo. The included methods are Modified Epley maneuver, Semont maneuver and Sham maneuver.

DETAILED DESCRIPTION:
This study was a prospective, double blinded, randomized, multicenter clinical trial. The enrolled posterior semicircular canal benign paroxysmal positional vertigo patients were randomized to one of the three treatment regimens when they are diagnosed with the Dix-Hallpike test. An then the patient was treated with one of the three maneuvers. After 20 minutes, the patient was examined with the Dix-Hallpike test again. The resolution of nystagmus and symptoms were checked. When the nystagmus was sustained, the same treatment was applied once again. And after 20 minutes, the patient was examined with the Dix-Hallpike test too. 1 day after and 7 days after, the patient was re-examined with the Dix-Hallpike test.

ELIGIBILITY:
Inclusion Criteria:

* a symptom of positional vertigo
* rotational and upbeating nystagmus in Dix-Hallpike test
* the nystagmus should be disappear within 60 seconds
* no spontaneous nystagmus

Exclusion Criteria:

* ages under 18 years
* suspicious or verified a central nervous system lesion
* traumatic vertigo patients
* other otologic disease(acute/chronic otitis media, otosclerosis, etc)
* other vestibular disease(vestibular neuronitis, Meniere's disease, etc)
* congenital nystagmus patients
* the patients with spinal disease
* the patients with the limitation of cervical movement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Initial Effectiveness of Treatment for the Posterior Semicircular Canal Benign Paroxysmal Positional Vertigo | 20 minutes
  The immediate effectiveness of treatment was determined by otolaryngologists with the Dix-Hallpike test 20 minutes after initial manerver applied. The investigator had no information of the treatment applied to the patient. The complete resolution means absence of nystagmus and paroxysmal vertigo symptom. If there was a sustained nystagmus, the latency and duration was measured.

SECONDARY OUTCOMES:
Delayed Effectiveness of Treatment for the Posterior Semicircular Canal Benign Paroxysmal Positional Vertigo | 1, 7 day
  Ather 1 day and 7 days after the initial treatment was applied, the patients were re-visit the clinic and re-examined with the Dix-Hallpike test. The absence of nystagmus and vertigo was determinded.

CONTACTS AND LOCATIONS:
Overall Officials: Hongju Park, Professor, Study Director — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea